CLINICAL TRIAL: NCT01932086
Title: A Randomized, Crossover Clinical Trial
Brief Title: Effects of White Rice, Brown Rice, and Black Rice on Postprandial Glucose and Lipid Profiles in Healthy Korean Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Director, Chonbuk National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTCF2_2011_RP_1
Record Dates: First submitted 2013-08-21; First posted 2013-08-30 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: male; Glucose; Triglyceride; Glycemic index; White rice; Brown rice; Black rice; Bread
MeSH Terms: interventions — Bread

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- White rice (Experimental)
  Interventions: Dietary Supplement: White rice diet; Dietary Supplement: Brown rice diet; Dietary Supplement: Black rice diet; Dietary Supplement: Bread; Other: Glucose solution
- Brown rice (Experimental)
  Interventions: Dietary Supplement: White rice diet; Dietary Supplement: Brown rice diet; Dietary Supplement: Black rice diet; Dietary Supplement: Bread; Other: Glucose solution
- Black rice (Experimental)
  Interventions: Dietary Supplement: White rice diet; Dietary Supplement: Brown rice diet; Dietary Supplement: Black rice diet; Dietary Supplement: Bread; Other: Glucose solution
- Bread (Active Comparator)
  Interventions: Dietary Supplement: White rice diet; Dietary Supplement: Brown rice diet; Dietary Supplement: Black rice diet; Dietary Supplement: Bread; Other: Glucose solution
- Glucose solution (Active Comparator)
  Interventions: Dietary Supplement: White rice diet; Dietary Supplement: Brown rice diet; Dietary Supplement: Black rice diet; Dietary Supplement: Bread

INTERVENTIONS:
Dietary Supplement: White rice diet — All test foods contained 50 g available carbohydrate from the test food products. A glass of 250 ml water was served together with the clinical trial food, and the participants were instructed to ingest the breakfast with 15 min
Dietary Supplement: Brown rice diet — All test foods contained 50 g available carbohydrate from the test food products. A glass of 250 ml water was served together with the clinical trial food, and the participants were instructed to ingest the breakfast with 15 min
Dietary Supplement: Black rice diet — All test foods contained 50 g available carbohydrate from the test food products. A glass of 250 ml water was served together with the clinical trial food, and the participants were instructed to ingest the breakfast with 15 min
Dietary Supplement: Bread — All test foods contained 50 g available carbohydrate from the test food products. A glass of 250 ml water was served together with the clinical trial food, and the participants were instructed to ingest the breakfast with 15 min
  Other Names: control diet
Other: Glucose solution — All test foods contained 50 g available carbohydrate from the test food products.and the participants were instructed to ingest the breakfast with 10 min.
  Other Names: Reference diet
  Arms: Black rice; Bread; Brown rice; White rice

SUMMARY:
This study was an open, 5-treatment, 5-sequence, 5-day cross-over randomized design clinical trial. The present study was carried out to compare the effects of white rice, brown rice, and black rice on postprandial glucose and lipid profiles in healthy human subjects, using a white bread as a positive control.

DETAILED DESCRIPTION:
After a 12-hour fast, oral glucose and meal tolerance was measured with blood samples drawn at times 0, 15, 30, 45, 60, 90, 120, 150 and 180 minutes and TG was at time 0, 1, 2, 3, 4, 5 and 6 hours.

1. Serum levels of glucose, insulin, and TG were analyzed by biochemical autoanalyzer. The area under the curve (AUC) changes in blood glucose, TG were computed by the trapezoidal method.
2. Glycemic index(GI): the area under the glucose response curve after consumption of a test food divided by the area under the curve after consumption of a control food containing the same amount of carbohydrate and calculated using 50 g glucose as the reference.

ELIGIBILITY:
Inclusion Criteria:

* Males, 19~60years old
* Bodyweight was more than 50 kg with ideal body weight within ±30%
* triglyceride (TG) levels less than 200 mg/dL
* Fasting blood glucose levels less than 100 mg/dL and an oral glucose tolerance test (OGTT) less than 140 mg/dL
* Able to give informed consent

Exclusion Criteria:

* Major medical illness such as cardiovascular, neurologic, psychiatric, renal, pulmonary and hepatic diseases
* History of disease that could interfere with the test products or impede their absorption such as gastrointestinal disease or gastrointestinal surgery
* Medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Poor vital sign (systolic blood pressure: below 100 mmHg or above 150 mmHg, diastolic blood pressure: below 65 mmHg or above95 mmHg)
* Allergic or hypersensitive to any of the ingredients in the test products; treated with any drug within past 2 weeks
* Participation in any other clinical trials within past 2 months
* Alcohol consumption above 21 units per week or abnormal screening laboratory test
* Being judged by the responsible physician of the local study center as unfit to participate in the study

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
1. Glucose, insulin AUC(incremental area under the curve) 2. Glycemic index(GI) | 2 hour postprandial blood glucose, insulin
  1. Plasma glucose and insulin will be measured at baseline, 15, 30, 45, 60, 90, 120, 180 and 240 minutes post ingestion of each test solution, and area under the curve will be calculated.
  2. Glycemic index (GI) was defined as the area under the glucose response curve after consumption of a test food divided by the area under the curve after consumption of a control food containing the same amount of carbohydrate and calculated using 50 g glucose as the reference. Plasma glucose will be measured at baseline, 15, 30, 45, 60, 90, and 120 minutes post ingestion of each test solution.
  GI= (incremental blood glucose area of test meal/incremental area of glucose) × 100

SECONDARY OUTCOMES:
Triglyceride iAUC(incremental area under the curve) | 6 hour postprandial blood triglyceride(TG)
  Triglyceride will be measured at baseline, 0, 1, 2, 3, 4, 5 and 6 hours post ingestion of each test solution, and area under the curve will be calculated.

OTHER OUTCOMES:
Homeostatic model assessment-insulin resistance(HOMA-IR), quantitative insulin sensitivity check index(QUICKI), Insulinogenic index(IGI) | fasting and postprandial (different times for 30min)
  1. HOMA-IR={fasting insulin(µU/㎖) x fasting glucose(m㏖/L)}/22.5
  2. QUICKI=1/log(insulin 0min)-log(glucose 0min)
  3. IGI=(insulin 30min-fasting insulin)/(glucose 30min-fasting glucose)

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Wan Chae, MD., PhD, Study Director — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea